CLINICAL TRIAL: NCT04551859
Title: Concordance of Pelvic Organ Mobility Measurements Between the Finite Element Model and the Dynamic Pelvic Floor MRI in Patients Undergoing a Sacrospinous Ligament Fixation Surgery
Brief Title: Concordance of Pelvic Organ Mobility Measurements Between the Finite Element Model and the Dynamic Pelvic Floor MRI in Patients Undergoing a Sacrospinofixation Surgery
Acronym: BiomécaRichter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020/510
Record Dates: First submitted 2020-09-07; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Sacrospinofixation; Apical Prolapse
Keywords: Sacrospinofixation; Prolapse; Richter; Vaginal vault; Sacrospinous ligament fixation
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacrospinofixation (Other): After accepting the surgeon's proposal to perform a sacrospinofixation to treat the pelvic organ prolapse, participation in this study will be proposed to the patient. It will not change the management or the course of the surgery
  Interventions: Other: Dynamic Pelvic Floor MRI

INTERVENTIONS:
Other: Dynamic Pelvic Floor MRI — 6 months after surgery, a Dynamic Pelvic Floor MRI is performed

SUMMARY:
The primary objective of this study is to demonstrate the feasibility of using a Finite Element model of pelvic organs by evaluating the concordance of pelvic organ mobility measurements performed by this mechanical model compared to the observations on the post-operative pelvic MRI in patients undergoing a sacrospinofixation surgery

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 80
* With at least a grade II apical prolapse according to the POP-Q classification
* Treated with a sacrospinous ligament fixation (SSF) by the vaginal route

Exclusion Criteria:

* History of abdominal, pelvic, vaginal or vulvar surgery except hysterectomy
* Association of another POP or urinary incontinence surgery (subvesical plication, levator myorrhaphy, plication of anterior rectal wall, perineorrhaphy ...)
* MRI contraindication
* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate with the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Concordance of mobility measurements of points C, Ba and Bp between the FE model and the dynamic MRI after SSF | 6 months after surgery
  Concordance of mobility measurements of the 3 points C, Ba, Bp during the defecation sequence, between the Finite Elements (FE) model and the dynamic pelvic floor MRI after sacrospinous ligament fixation (SSF)

SECONDARY OUTCOMES:
Concordance of mobility measurements of points Aa and Ap between the FE model and the dynamic MRI after SSF | 6 months after surgery
  Concordance of mobility measurements of points Aa and Ap during the defecation sequence, between the Finite Elements (FE) model and the dynamic pelvic floor MRI after sacrospinous ligament fixation SSF)
Comparison of the pelvic organ mobility before and after surgery | 6 months after surgery
  Comparison of the mobility of the different points of the POP-Q classification (C, Ba, Bp, Aa, Ap) before and after surgery
Elasticity study of the vaginal tissue (Lille) | after surgery (day 0)
  Elasticity study of the vaginal tissue removed during surgery (for patients operated in Lille only)
Concordance of mobility measurements between FE model enhanced by the vaginal tissue analysis and the dynamic MRI after SSF | 6 months after surgery
  Concordance of mobility measurements of the POP-Q points (C, Ba, Bp, Aa, Ba) during the defecation sequence, between the Finite Elements (FE) model enhanced by the analysis of the vaginal tissue sampling and the dynamic pelvic floor MRI after sacrospinous ligament fixation (SSF)

REFERENCES:
- [Background] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Background] de Tayrac R, Letouzey V, Costa P, Haab F, Delmas V. [Treatment of uterine prolapse and vaginal vault by vaginal route]. Prog Urol. 2009 Dec;19(13):1074-9. doi: 10.1016/j.purol.2009.09.025. Epub 2009 Oct 21. French. PMID 19969278
- [Background] Cosson M, Rubod C, Vallet A, Witz JF, Dubois P, Brieu M. Simulation of normal pelvic mobilities in building an MRI-validated biomechanical model. Int Urogynecol J. 2013 Jan;24(1):105-12. doi: 10.1007/s00192-012-1842-8. Epub 2012 Jun 16. PMID 22707008
- [Background] Lamblin G, Mayeur O, Giraudet G, Jean Dit Gautier E, Chene G, Brieu M, Rubod C, Cosson M. Pathophysiological aspects of cystocele with a 3D finite elements model. Arch Gynecol Obstet. 2016 Nov;294(5):983-989. doi: 10.1007/s00404-016-4150-6. Epub 2016 Jul 11. PMID 27402504
- [Background] Jeanditgautier E, Mayeur O, Brieu M, Lamblin G, Rubod C, Cosson M. Mobility and stress analysis of different surgical simulations during a sacral colpopexy, using a finite element model of the pelvic system. Int Urogynecol J. 2016 Jun;27(6):951-7. doi: 10.1007/s00192-015-2917-0. Epub 2016 Jan 11. PMID 26755057
- [Background] Cosson M, Rubod C, Vallet A, Witz JF, Brieu M. [Biomechanical modeling of pelvic organ mobility: towards personalized medicine]. Bull Acad Natl Med. 2011 Nov;195(8):1869-83; discussion 1883. French. PMID 22844748
- [Background] Estrade JP, Agostini A, Roger V, Dallay D, Blanc B, Cravello L. [Posthysterectomy prolapse: results of sacrospinous ligament fixation]. J Gynecol Obstet Biol Reprod (Paris). 2005 Sep;34(5):481-7. doi: 10.1016/s0368-2315(05)82856-x. French. PMID 16142139
- [Background] Maher C, Feiner B, Baessler K, Christmann-Schmid C, Haya N, Brown J. Surgery for women with apical vaginal prolapse. Cochrane Database Syst Rev. 2016 Oct 1;10(10):CD012376. doi: 10.1002/14651858.CD012376. PMID 27696355
- [Derived] Lallemant M, Shimojyo AA, Mayeur O, Ramanah R, Rubod C, Kerbage Y, Cosson M. Mobility analysis of a posterior sacrospinous fixation using a finite element model of the pelvic system. PLoS One. 2024 Mar 21;19(3):e0299012. doi: 10.1371/journal.pone.0299012. eCollection 2024. PMID 38512958